CLINICAL TRIAL: NCT06632301
Title: DEXA Bone Density Analysis to Analyze the Loading Concept of the CoreHip® Prosthesis
Brief Title: DEXA Bone Density Analysis of the CoreHip® Prosthesis System
Acronym: CODEX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAG-G-H-23009
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Primary Osteoarthritis; Cartilage Degeneration; Osteoarthritis, Hip; Inflammatory Arthritis; Osteonecrosis of Femoral Head; Traumatic Disorder
Keywords: Total Hip Arthroplasty; DEXA Bone Density Analysis
MeSH Terms: conditions — Osteoarthritis, Hip; Arthritis; Femur Head Necrosis; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DEXA (Experimental): DEXA bone density analysis to analyze the loading concept of the CoreHip® Prosthesis System
  Interventions: Device: Primary hip replacement with cementless stem

INTERVENTIONS:
Device: Primary hip replacement with cementless stem — Total Hip Arthroplasty is today one of the most established surgical orthopaedic procedures worldwide.

SUMMARY:
The goal of this interventional post-market follow-up study is to evaluate radiological changes in the diaphyseal bone density (Gruen Zones 3 and 4) within 24 months postoperative in patients treated with CoreHip® primary cementless stem. The DEXA bone density analysis is used.

DETAILED DESCRIPTION:
Additional diagnostic examination: DEXA-Analysis. A DEXA scan is an imaging test that measures bone density (strength). The results can provide helpful details about risk for osteoporosis (bone loss) and fractures. Furthermore we would like to find out more about stress shielding processes around our prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral hip osteoarthritis
* Indication for CoreHip Standard hip stem according to preoperative planning
* Written Informed Consent
* Age 35-85 years
* According to the assessment of the study doctor, the patient is therapy compliant and able to attend the follow-up visits

Exclusion Criteria:

* Femoral neck fractures
* Pregnancy
* BMI > 35
* History of femoral fracture or previous surgery on the same hip
* Metabolic bone disease, use of steroids or other drugs affecting bone metabolism
* Intraoperative bone cracks
* Severe osteoarthritis of the contralateral hip
* THA of the contralateral side or other event leading to restricted weight bearing during the study period

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Radiological changes in the diaphyseal bone density (Gruen Zones 3 and 4) | within 24 months postoperative
  Changes in bone mineral density (BMD) according to Gruen.

SECONDARY OUTCOMES:
Clinical Results: Joint Function (Harris Hip Score) | preoperative, at discharge (1 week postop) and 12 months postoperative
  The functional results of the operated hip will be assessed with the Harris Hip Score (HHS) and evaluated over time.
Development of Quality of Life (EQ-5D-5L) | preoperative, at discharge (1 week postop) and 12 months postoperative
  The EQ-5D-5L score is a generic score used to document the well-being of the patient.
Development of Forgotten Joint Score | preoperative, at discharge (1 week postop) and 12 months postoperative
  The EQ-5D-5L score is a generic score used to document the well-being of the patient.
Development of Pain | preoperative, at discharge (1 week postop) and 12 months postoperative
  The development of pain is measured with the Visual analog scale [VAS] a measure of pain intensity. The scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [on 100-mm scale].
Development of Pain | preoperative, at discharge (1 week postop) and 12 months postoperative
  Radiological changes in the diaphyseal bone density (DEXA BMD progression over time in all Gruen Zones (Zone 1-7)

CONTACTS AND LOCATIONS:
Overall Officials: Henning Windhagen, Prof. Dr., Principal Investigator — Orthopädische Kliniken im Annastift, MHH
Locations (1):
- Medizinische Hochschule Hannover, Hanover, Germany